CLINICAL TRIAL: NCT03754556
Title: Study on the Association of Uterine Perforation and Intrauterine Device (IUD) Expulsion With Breastfeeding Status at the Time of IUD Insertion and Postpartum Timing of IUD Insertion in Electronic Medical Record Databases - A Postmarketing Requirement for Mirena
Brief Title: Study on Medical Records of Women Using an Intrauterine Device (IUD) to Analyze the Risks That the IUD Will be Expelled or Perforates the Womb in Relation to Breastfeeding, the Point in Time When the IUD Was Inserted After Childbirth and in Relation to Different Types of IUDs
Acronym: APEX IUD
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19682
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Intrauterine Devices
Keywords: Contraception; Breast-feeding; Electronic medical records; Uterine perforation; Expulsion of intrauterine device
MeSH Terms: conditions — Breast Feeding; Uterine Perforation | interventions — Intrauterine Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with IUD: Women with an intrauterine device (IUD) and electronic health records in the Kaiser Permanente Northern California (KPNC), Kaiser Permanente Southern California (KPSC), Kaiser Permanente Washington (KPWA) and the Regenstrief Institute (RI) databases.
  Interventions: Device: Intrauterine device

INTERVENTIONS:
Device: Intrauterine device — Intrauterine devices, e.g. BAY86-5028 (Mirena, Skyla, Kyleena), Liletta and ParaGard
  Other Names: Levonorgestrel, Copper IUD

SUMMARY:
Study to analyze electronic medical records of women using an intrauterine device (IUD). The study was required by the FDA for the marketed IUD Mirena (US Post-marketing requirement; short name of study: APEX IUD).

The study analyzed the risks that the IUD was expelled or perforated the womb for the following group comparisons:

* Women who were breastfeeding at the time of IUD insertion and within 52 weeks postpartum versus women who were not breastfeeding at the time of IUD insertion and within 52 weeks postpartum.
* Women who had a first observed IUD insertion within different time periods after childbirth (i.e., ≤ 6 weeks, > 6 weeks and ≤ 14 weeks, > 14 weeks and ≤ 52 weeks) versus women who had their first observed IUD insertion more than 52 weeks after childbirth, including women without a recorded delivery within the past 52 weeks. An additional analysis involved 5-level postpartum timing (i.e., 0 to 3 days, 4 days to ≤ 6 weeks, > 6 weeks to ≤ 14 weeks, > 14 weeks to ≤ 52 weeks) versus the > 52 week postpartum group.

The study also analyzed the risks that the IUD was expelled or perforated the womb for different types of IUDs. In addition, the study aimed to assess the following interactions:

* The extent to which the type of IUD (IUDs releasing the hormone LNG versus Copper IUDs) modified the risk that an IUD was expelled or perforated the womb in relation to breastfeeding and/ or in relation to the point in time when the IUD was inserted after childbirth.
* The extent to which the breastfeeding status modified the risk that an IUD was expelled or perforated the womb in relation to the point in time when the IUD was inserted after childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Women with evidence in the database of insertion of an IUD (e.g. levonorgestrel-releasing, copper) during the study time window for each site
* Enrolled in the database with electronic medical records available for review for at least 12 months before the IUD insertion

Exclusion Criteria:

- Women with more than 50 years of age at the time of the IUD-insertion

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women with IUD-insertion
Sampling Method: Non-Probability Sample
Enrollment: 326658 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Kaiser Permanente Northern California, Oakland, California
  - Kaiser Permanente Southern California, Pasadena, California
  - Regenstrief Institute, Indianapolis, Indiana
  - Kaiser Permanente Washington, Seattle, Washington

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a retrospective cohort study, using the data from three health care systems: Kaiser Permanente Northern California (KPNC), Kaiser Permanente Southern California (KPSC), Kaiser Permanente Washington (KPWA) and one research institute with access to a health information exchange, Regenstrief Institute (RI)
Pre-assignment Details: Between 01 January 2001 and 30 April 2018, 326658 participants were identified: 322898 participants with intrauterine device (IUD) type available and 94817 participants with breastfeeding status available (and IUD insertion within 12 months postpartum)
Period: Overall Study
Arm/Group | Women With IUD
Started | 326658
Completed | 326658
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
Age, Customized [Count of Participants; unit: Participants]
  ≤ 28 years | 119469
  > 28 to ≤ 36 years | 107871
  > 36 to ≤ 50 years | 99318
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 326658
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 38911
  Hispanic black | 696
  Hispanic white | 42501
  Hispanic other | 56180
  Non-Hispanic black | 28323
  Non-Hispanic white | 137102
  Other or multiple | 16357
  Unknown | 6588
Breastfeeding status [Count of Participants; unit: Participants]
  Yes (for those ≤ 52 weeks postpartum) | 64186
  No (for those ≤ 52 weeks postpartum) | 30631
  Undetermined (for those ≤ 52 weeks postpartum) | 3007
  No delivery in the past year | 228834
Postpartum time of IUD insertion [Count of Participants; unit: Participants]
  0 to 3 days | 2788
  4 days to ≤ 6 weeks | 17272
  > 6 to ≤ 14 weeks | 56047
  > 14 to ≤ 52 weeks | 21717
  > 52 weeks or no delivery | 228834
Menorrhagia [Count of Participants; unit: Participants]
  ≤ 12 months before insertion | 32552
  > 12 months or no diagnosis | 294106
IUD type [Count of Participants; unit: Participants]
  Levonorgestrel (LNG)-IUD | 259234
  Copper IUD | 63664
  Unknown | 3760

OUTCOME MEASURES:

1. Primary Outcome: Crude Incidence Rate of Uterine Perforation Stratified by Breastfeeding Status Among Women Within 52 Weeks Postpartum-first Observed IUD Insertions
Description: Crude incidence rate was calculated as the number of outcomes occurring during the person-time at risk divided by the total person-time at risk (in person-years)
Time Frame: Up to 11 years
Population: Women who were within 52 weeks postpartum and were or were not breastfeeding at the time of IUD insertion
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 94817
per 1000 person-years
  Breastfeeding: number analyzed (Participants) | 64186
  Breastfeeding | 4.25 [3.89 to 4.62]
  Not breastfeeding: number analyzed (Participants) | 30631
  Not breastfeeding | 2.50 [2.11 to 2.94]

2. Primary Outcome: Cumulative Incidence of Uterine Perforation Stratified by Breastfeeding Status Among Women Within 52 Weeks Postpartum-first Observed IUD Insertions
Description: Crude estimates of the cumulative incidence, defined as number of outcomes occurring up to a time point out of the number of IUD insertions
Time Frame: At 1 year and 5 years of follow-up
Population: Women who were within 52 weeks postpartum and were or were not breastfeeding at the time of IUD insertion
Measure: Number (95% Confidence Interval); unit: number of outcomes/IUD insertions (%)
Arm/Group | Women With IUD
Number analyzed (Participants) | 94817
number of outcomes/IUD insertions (%)
  Breastfeeding, 1 year of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 1 year of follow-up | 0.60 [0.54 to 0.67]
  Not breastfeeding, 1 year of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 1 year of follow-up | 0.35 [0.29 to 0.43]
  Breastfeeding, 5 years of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 5 years of follow-up | 1.61 [1.43 to 1.81]
  Not breastfeeding, 5 years of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 5 years of follow-up | 0.88 [0.71 to 1.08]

3. Primary Outcome: Adjusted Hazard Ratio (HR) for Breastfeeding Status and Uterine Perforation-first Observed IUD Insertions
Description: Propensity score-adjusted hazard ratio to evaluate whether the risk of uterine perforation among women who were breastfeeding at the time of first observed IUD insertion differs from the risk of uterine perforation among women who were not breastfeeding at the time of first observed IUD insertion
Time Frame: Up to 11 years
Population: Women who had given birth in the previous 52 weeks and had breastfeeding status "yes" or "no" were included in this analysis
Measure: Number (95% Confidence Interval); unit: ajusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 94817
ajusted hazard ratio | 1.37 [1.12 to 1.66]

4. Primary Outcome: Crude Incidence Rate of Uterine Perforation Categorized by Postpartum Timing-first Observed IUD Insertions
Description: as for outcome 1
Time Frame: Up to 11 years
Population: Women with first observed IUD insertions at different postpartum timing or women without recorded delivery within the past 52 weeks
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
per 1000 person-years
  ≤ 6 weeks postpartum: number analyzed (Participants) | 20060
  ≤ 6 weeks postpartum | 5.14 [4.44 to 5.92]
  > 6 weeks and ≤ 14 weeks postpartum: number analyzed (Participants) | 56047
  > 6 weeks and ≤ 14 weeks postpartum | 3.77 [3.42 to 4.15]
  > 14 weeks and ≤ 52 weeks postpartum: number analyzed (Participants) | 21717
  > 14 weeks and ≤ 52 weeks postpartum | 2.24 [1.80 to 2.75]
  > 52 weeks postpartum or no delivery: number analyzed (Participants) | 228834
  > 52 weeks postpartum or no delivery | 0.68 [0.61 to 0.76]

5. Primary Outcome: Cumulative Incidence of Uterine Perforation Categorized by Postpartum Timing-first Observed IUD Insertions
Description: as for outcome 2
Time Frame: At 1 year and 5 years of follow-up
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: number of outcomes/IUD insertions (%)
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
number of outcomes/IUD insertions (%)
  ≤ 6 weeks postpartum (pp), 1 year of follow-up: number analyzed (Participants) | 20060
  ≤ 6 weeks postpartum (pp), 1 year of follow-up | 0.70 [0.59 to 0.84]
  > 6 weeks and ≤ 14 weeks pp, 1 year of follow-up: number analyzed (Participants) | 56047
  > 6 weeks and ≤ 14 weeks pp, 1 year of follow-up | 0.54 [0.48 to 0.61]
  > 14 weeks and ≤ 52 weeks pp, 1 year of follow-up: number analyzed (Participants) | 21717
  > 14 weeks and ≤ 52 weeks pp, 1 year of follow-up | 0.33 [0.26 to 0.43]
  > 52 weeks pp or no delivery, 1 year of follow-up: number analyzed (Participants) | 228834
  > 52 weeks pp or no delivery, 1 year of follow-up | 0.07 [0.06 to 0.08]
  ≤ 6 weeks pp, 5 years of follow-up: number analyzed (Participants) | 20060
  ≤ 6 weeks pp, 5 years of follow-up | 1.89 [1.55 to 2.31]
  > 6 weeks and ≤ 14 weeks pp, 5 years of follow-up: number analyzed (Participants) | 56047
  > 6 weeks and ≤ 14 weeks pp, 5 years of follow-up | 1.42 [1.25 to 1.61]
  > 14 weeks and ≤ 52 weeks pp, 5 years of follow-up: number analyzed (Participants) | 21717
  > 14 weeks and ≤ 52 weeks pp, 5 years of follow-up | 0.74 [0.57 to 0.97]
  > 52 weeks pp or no delivery, 5 years of follow-up: number analyzed (Participants) | 228834
  > 52 weeks pp or no delivery, 5 years of follow-up | 0.29 [0.26 to 0.34]

6. Primary Outcome: Adjusted Hazard Ratio (HR) for Postpartum Timing and Uterine Perforation-first Observed IUD Insertions
Description: Adjusted for propensity scores and breastfeeding status, to evaluate whether the risk of uterine perforation among women who had a first observed IUD insertion within different time periods postpartum differs from the risk of uterine perforation among women who had their first observed IUD insertion more than 52 weeks postpartum, including women without a recorded delivery within the past 52 weeks. Reference group: IUD insertion > 52 weeks postpartum
Time Frame: Up to 11 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: ajusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
ajusted hazard ratio
  ≤ 6 weeks postpartum: number analyzed (Participants) | 20060
  ≤ 6 weeks postpartum | 6.29 [4.50 to 8.79]
  > 6 weeks and ≤ 14 weeks postpartum: number analyzed (Participants) | 56047
  > 6 weeks and ≤ 14 weeks postpartum | 4.65 [3.49 to 6.20]
  > 14 weeks and ≤ 52 weeks postpartum: number analyzed (Participants) | 21717
  > 14 weeks and ≤ 52 weeks postpartum | 2.94 [2.16 to 4.01]

7. Primary Outcome: Adjusted Hazard Ratio (HR) for Postpartum Timing Risk 14-week Cut Point and Uterine Perforation-first Observed IUD Insertions
Description: Adjusted for propensity scores and breastfeeding status, to estimate the risk of uterine perforation among women who had a first observed IUD insertion early in the postpartum period (i.e., up to 14 weeks postpartum) versus those who had a first observed IUD insertion late in the postpartum period (i.e., more than 14 weeks postpartum, including women without recorded delivery within the past 52 weeks). Reference group: IUD insertion >14 weeks postpartum or with no recorded delivery
Time Frame: Up to 11 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted hazard ratio | 3.44 [2.70 to 4.40]

8. Primary Outcome: Adjusted Hazard Ratio (HR) for Postpartum Timing Risk 36-week Cut Point and Uterine Perforation-first Observed IUD Insertions
Description: Adjusted for propensity scores and breastfeeding status, to estimate the risk of uterine perforation among women who had a first observed IUD insertion ≤ 36 weeks postpartum versus women who had a first observed IUD insertion > 36 weeks postpartum, including women without recorded delivery within the past 52 weeks. Reference group: IUD insertion >36 weeks postpartum or with no recorded delivery
Time Frame: Up to 11 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted hazard ratio | 4.36 [3.45 to 5.51]

9. Primary Outcome: Adjusted Incidence Rate Ratio (IRR) for Uterine Perforation-first Observed IUD Insertions
Description: Adjusted for propensity score, overall and stratified by breastfeeding status at the time of IUD insertion for ≤ 36 weeks postpartum at IUD insertion versus > 36 weeks postpartum or with no recorded delivery, at 1 year and 5 years of follow-up. Reference group: > 36 weeks or no delivery
Time Frame: At 1 year and 5 years of follow-up
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: adjusted incidence rate ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted incidence rate ratio
  Overall, 1 year of follow-up | 4.72 [3.74 to 5.96]
  Overall, 5 years of follow-up | 4.10 [3.43 to 4.90]
  Breastfeeding, 1 year of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 1 year of follow-up | 1.11 [0.57 to 2.47]
  Not breastfeeding, 1 year of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 1 year of follow-up | 6.61 [5.03 to 8.76]
  Breastfeeding, 5 years of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 5 years of follow-up | 1.47 [0.80 to 3.07]
  Not breastfeeding, 5 years of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 5 years of follow-up | 4.86 [4.00 to 5.93]

10. Primary Outcome: Adjusted Incidence Rate Difference (IRD) for Uterine Perforation-first Observed IUD Insertions
Description: Propensity score-adjusted incidence rate differences (per 1,000 person-years) for uterine perforation for women ≤ 36 weeks postpartum at IUD insertion compared with those who were > 36 weeks postpartum or with no recorded delivery, 1 year of follow-up and 5 years of follow-up, overall and stratified by breastfeeding status. Reference group: > 36 weeks or no delivery
Time Frame: At 1 year and 5 years of follow-up
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
per 1000 person-years
  Overall, 1 year of follow-up | 3.75 [3.05 to 4.45]
  Overall, 5 years of follow-up | 2.28 [1.93 to 2.63]
  Breastfeeding, 1 year of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 1 year of follow-up | 0.63 [-3.39 to 4.64]
  Not breastfeeding, 1 year of follow-up: number analyzed (Participants) | 64186
  Not breastfeeding, 1 year of follow-up | 3.92 [3.22 to 4.63]
  Breastfeeding, 5 years of follow-up: number analyzed (Participants) | 30631
  Breastfeeding, 5 years of follow-up | 1.38 [-0.46 to 3.21]
  Not breastfeeding, 5 years of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 5 years of follow-up | 2.33 [1.97 to 2.69]

11. Primary Outcome: Crude Incidence Rate of Uterine Perforation Stratified by IUD Type-first Observed IUD Insertions
Description: as for outcome 1
Time Frame: Up to 11 years
Population: Women with either LNG-IUD (levonorgestrel-releasing intrauterine system) or copper IUD insertions
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 322898
per 1000 person-years
  LNG-IUD: number analyzed (Participants) | 259534
  LNG-IUD | 1.64 [1.53 to 1.76]
  Copper IUD: number analyzed (Participants) | 63664
  Copper IUD | 1.27 [1.08 to 1.48]

12. Primary Outcome: Cumulative Incidence of Uterine Perforation Stratified by IUD Type-first Observed IUD Insertions
Description: as for outcome 2
Time Frame: At 1 year and 5 years of follow-up
Population: Women with either LNG-IUD (levonorgestrel-releasing intrauterine system) or copper IUD insertions
Measure: Number (95% Confidence Interval); unit: number of outcomes/IUD insertions (%)
Arm/Group | Women With IUD
Number analyzed (Participants) | 322898
number of outcomes/IUD insertions (%)
  LNG-IUD, 1 year of follow up: number analyzed (Participants) | 259234
  LNG-IUD, 1 year of follow up | 0.22 [0.20 to 0.24]
  Copper IUD, 1 year of follow up: number analyzed (Participants) | 63664
  Copper IUD, 1 year of follow up | 0.16 [0.13 to 0.20]
  LNG-IUD, 5 years of follow up: number analyzed (Participants) | 259234
  LNG-IUD, 5 years of follow up | 0.63 [0.57 to 0.68]
  Copper IUD, 5 years of follow up: number analyzed (Participants) | 63664
  Copper IUD, 5 years of follow up | 0.55 [0.44 to 0.68]

13. Primary Outcome: Adjusted Hazard Ratio (HR) for IUD Type and Uterine Perforation-first Observed IUD Insertions
Description: Propensity score-adjusted hazard ratio to evaluate whether the risk of uterine perforation among women with LNG-releasing IUD at the time of first observed IUD insertion differs from the risk of uterine perforation among women with copper IUD at the time of first observed IUD insertion
Time Frame: Up to 11 years
Population: Women with either LNG-IUD (levonorgestrel-releasing intrauterine system) or copper IUD insertions
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 322898
adjusted hazard ratio | 1.49 [1.25 to 1.78]

14. Primary Outcome: Crude Incidence Rate of Uterine Perforation Stratified by Menorrhagia Status-first Observed IUD Insertions
Description: as for outcome 1
Time Frame: Up to 11 years
Population: Women with menorrhagia (heavy menstrual bleeding) status (yes/no) in the 12 months before IUD insertion
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
per 1000 person-years
  Yes: number analyzed (Participants) | 32552
  Yes | 1.00 [0.77 to 1.28]
  No: number analyzed (Participants) | 294106
  No | 1.63 [1.53 to 1.74]

15. Primary Outcome: Cumulative Incidence of Uterine Perforation Stratified by Menorrhagia Status-first Observed IUD Insertions
Description: as for outcome 2
Time Frame: At 1 year and 5 years of follow-up
Population: Women with menorrhagia (heavy menstrual bleeding) status (yes/no) in the 12 months before IUD insertion
Measure: Number (95% Confidence Interval); unit: number of outcomes/IUD insertions (%)
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
number of outcomes/IUD insertions (%)
  Yes, 1 year of follow-up: number analyzed (Participants) | 32552
  Yes, 1 year of follow-up | 0.10 [0.07 to 0.14]
  No, 1 year of follow-up: number analyzed (Participants) | 294106
  No, 1 year of follow-up | 0.22 [0.20 to 0.24]
  Yes, 5 years of follow-up: number analyzed (Participants) | 32552
  Yes, 5 years of follow-up | 0.41 [0.31 to 0.56]
  No, 5 years of follow-up | 0.63 [0.58 to 0.69]

16. Primary Outcome: Adjusted Hazard Ratio (HR) for Menorrhagia Status and Uterine Perforation-first Observed IUD Insertions
Description: Propensity score-adjusted hazard ratio to evaluate whether the risk of uterine perforation among women using an IUD who have at least one diagnosis code indicating menorrhagia in the 12 months before IUD insertion differs from the risk of uterine perforation among women who do not have this indication
Time Frame: Up to 11 years
Population: Women with menorrhagia (heavy menstrual bleeding) status (yes/no) in the 12 months before IUD insertion
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted hazard ratio | 1.38 [1.01 to 1.88]

17. Primary Outcome: Effect Modification of Breastfeeding Status on Postpartum Timing for Uterine Perforation
Description: Propensity score-adjusted hazard ratios to evaluate the extent to which breastfeeding status (yes vs. no) modified the association of uterine perforation for women with IUD insertion at different time periods postpartum (i.e., IUD insertion ≤ 14 weeks versus IUD insertion > 14 weeks postpartum) among women with a recorded delivery within the past 52 weeks at the time of the first observed IUD insertion
Time Frame: Up to 11 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 94817
adjusted hazard ratio
  ≤ 14 weeks, breastfeeding yes vs.no | 1.28 [1.02 to 1.61]
  > 14 to ≤ 52 weeks, breastfeeding yes vs.no | 2.41 [1.47 to 3.95]
  Breastfeeding yes, ≤ 14 vs. > 14 to ≤ 52 weeks: number analyzed (Participants) | 64186
  Breastfeeding yes, ≤ 14 vs. > 14 to ≤ 52 weeks | 1.36 [1.01 to 1.83]
  Breastfeeding no, ≤ 14 vs. > 14 to ≤ 52 weeks: number analyzed (Participants) | 30631
  Breastfeeding no, ≤ 14 vs. > 14 to ≤ 52 weeks | 2.56 [1.62 to 4.02]

18. Primary Outcome: Effect Modification of IUD Type on Breastfeeding Status for Uterine Perforation
Description: Propensity score-adjusted hazard ratios to evaluate the extent to which type of IUD (LNG-IUD vs. copper IUD) modified the association between uterine perforation and breastfeeding among women who were and were not breastfeeding at the time of first observed IUD insertion
Time Frame: Up to 11 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 94205
adjusted hazard ratio
  LNG-IUD, breastfeeding yes vs.no: number analyzed (Participants) | 72201
  LNG-IUD, breastfeeding yes vs.no | 1.33 [1.07 to 1.64]
  Copper IUD, breastfeeding yes vs.no: number analyzed (Participants) | 22004
  Copper IUD, breastfeeding yes vs.no | 1.66 [0.94 to 2.94]

19. Primary Outcome: Effect Modification of IUD Type on Postpartum Timing for Uterine Perforation
Description: Adjusted for propensity score and breastfeeding status, to evaluate the extent to which type of IUD (LNG-IUD vs. copper IUD) modified the association between uterine perforation and postpartum timing of IUD insertion for women with IUD insertion at different time periods postpartum (i.e., ≤ 6 weeks, > 6 and ≤ 14 weeks, > 14 and ≤ 52 weeks) versus IUD insertion more than 52 weeks postpartum, including no recorded delivery within the past 52 weeks, at the time of the first observed IUD insertion. Reference group: LNG-IUD or Copper IUD, > 52 weeks or no delivery
Time Frame: Up to 11 years
Population: Women with either LNG-IUD (levonorgestrel-releasing intrauterine system) or copper IUD insertions
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 322898
adjusted hazard ratio
  LNG-IUD, ≤ 6 weeks: number analyzed (Participants) | 15631
  LNG-IUD, ≤ 6 weeks | 6.78 [4.74 to 9.70]
  LNG-IUD, > 6 to ≤ 14 weeks: number analyzed (Participants) | 42760
  LNG-IUD, > 6 to ≤ 14 weeks | 5.11 [3.75 to 6.95]
  LNG-IUD, > 14 to ≤ 52 weeks: number analyzed (Participants) | 16110
  LNG-IUD, > 14 to ≤ 52 weeks | 3.13 [2.21 to 4.42]
  Copper IUD, ≤ 6 weeks: number analyzed (Participants) | 4228
  Copper IUD, ≤ 6 weeks | 4.30 [2.38 to 7.75]
  Copper IUD, > 6 to ≤ 14 weeks: number analyzed (Participants) | 12934
  Copper IUD, > 6 to ≤ 14 weeks | 2.61 [1.56 to 4.36]
  Copper IUD, > 14 to ≤ 52 weeks: number analyzed (Participants) | 5379
  Copper IUD, > 14 to ≤ 52 weeks | 2.01 [1.05 to 3.85]

20. Secondary Outcome: Crude Incidence Rate of IUD Expulsion Stratified by Breastfeeding Status Among Women Within 52 Weeks Postpartum-first Observed IUD Insertions
Description: as for outcome 1
Time Frame: Up to 11 years
Population: Women who were within 52 weeks postpartum and were or were not breastfeeding at the time of IUD insertion
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 94817
per 1000 person-years
  Breastfeeding: number analyzed (Participants) | 64186
  Breastfeeding | 10.23 [9.68 to 10.81]
  Not breastfeeding: number analyzed (Participants) | 30631
  Not breastfeeding | 14.58 [13.62 to 15.59]

21. Secondary Outcome: Cumulative Incidence of IUD Expulsion Stratified by Breastfeeding Status Among Women Within 52 Weeks Postpartum-first Observed IUD Insertions
Description: as for outcome 2
Time Frame: At 1 year and 5 years of follow-up
Population: Women who were within 52 weeks postpartum and were or were not breastfeeding at the time of IUD insertion
Measure: Number (95% Confidence Interval); unit: number of outcomes/IUD insertions (%)
Arm/Group | Women With IUD
Number analyzed (Participants) | 94817
number of outcomes/IUD insertions (%)
  Breastfeeding, 1 year of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 1 year of follow-up | 1.55 [1.44 to 1.65]
  Not breastfeeding, 1 year of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 1 year of follow-up | 2.45 [2.27 to 2.65]
  Breastfeeding, 5 years of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 5 years of follow-up | 3.49 [3.25 to 3.73]
  Not breastfeeding, 5 years of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 5 years of follow-up | 4.57 [4.22 to 4.95]

22. Secondary Outcome: Adjusted Hazard Ratio (HR) for Breastfeeding Status and IUD Expulsion-first Observed IUD Insertions
Description: Propensity score-adjusted to evaluate whether the risk of IUD expulsion among women who were breastfeeding at the time of first observed IUD insertion differs from the risk of IUD expulsion among women who were not breastfeeding at the time of first observed IUD insertion
Time Frame: Up to 11 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 94817
adjusted hazard ratio | 0.71 [0.64 to 0.78]

23. Secondary Outcome: Crude Incidence Rate of IUD Expulsion Categorized by Postpartum Timing-first Observed IUD Insertions
Description: as for outcome 1
Time Frame: Up to 11 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
per 1000 person-years
  ≤ 3 days: number analyzed (Participants) | 2788
  ≤ 3 days | 46.54 [40.54 to 53.18]
  4 days to ≤ 6 weeks: number analyzed (Participants) | 17272
  4 days to ≤ 6 weeks | 10.88 [9.78 to 12.08]
  ≤ 6 weeks postpartum: number analyzed (Participants) | 20060
  ≤ 6 weeks postpartum | 15.33 [14.10 to 16.65]
  > 6 weeks and ≤ 14 weeks postpartum: number analyzed (Participants) | 56047
  > 6 weeks and ≤ 14 weeks postpartum | 9.29 [8.73 to 9.87]
  > 14 weeks and ≤ 52 weeks postpartum: number analyzed (Participants) | 21717
  > 14 weeks and ≤ 52 weeks postpartum | 14.36 [13.22 to 15.57]
  > 52 weeks postpartum or no delivery: number analyzed (Participants) | 228834
  > 52 weeks postpartum or no delivery | 14.93 [14.57 to 15.29]

24. Secondary Outcome: Cumulative Incidence of IUD Expulsion Categorized by Postpartum Timing-first Observed IUD Insertions
Description: as for outcome 2
Time Frame: At 1 year and 5 years of follow-up
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: number of outcomes/IUD insertions (%)
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
number of outcomes/IUD insertions (%)
  ≤ 3 days, 1 year of follow-up: number analyzed (Participants) | 2788
  ≤ 3 days, 1 year of follow-up | 7.84 [6.83 to 9.00]
  4 days to ≤ 6 weeks, 5 years of follow-up: number analyzed (Participants) | 17272
  4 days to ≤ 6 weeks, 5 years of follow-up | 3.87 [3.40 to 4.42]
  ≤ 6 weeks postpartum (pp), 1 year of follow-up: number analyzed (Participants) | 20060
  ≤ 6 weeks postpartum (pp), 1 year of follow-up | 2.46 [2.24 to 2.71]
  > 6 weeks and ≤ 14 weeks pp, 1 year of follow-up: number analyzed (Participants) | 56047
  > 6 weeks and ≤ 14 weeks pp, 1 year of follow-up | 1.40 [1.30 to 1.51]
  > 14 weeks and ≤ 52 weeks pp, 1 year of follow-up: number analyzed (Participants) | 21717
  > 14 weeks and ≤ 52 weeks pp, 1 year of follow-up | 2.33 [2.12 to 2.56]
  > 52 weeks pp or no delivery, 1 year of follow-up: number analyzed (Participants) | 228834
  > 52 weeks pp or no delivery, 1 year of follow-up | 2.49 [2.42 to 2.56]
  ≤ 3 days, 5 years of follow-up: number analyzed (Participants) | 2788
  ≤ 3 days, 5 years of follow-up | 10.73 [9.12 to 12.61]
  4 days to ≤ 6 weeks, 1 year of follow-up: number analyzed (Participants) | 17272
  4 days to ≤ 6 weeks, 1 year of follow-up | 1.61 [1.42 to 1.84]
  ≤ 6 weeks pp, 5 years of follow-up: number analyzed (Participants) | 20060
  ≤ 6 weeks pp, 5 years of follow-up | 4.81 [4.33 to 5.33]
  > 6 weeks and ≤ 14 weeks pp, 5 years of follow-up: number analyzed (Participants) | 56047
  > 6 weeks and ≤ 14 weeks pp, 5 years of follow-up | 3.18 [2.95 to 3.42]
  > 14 weeks and ≤ 52 weeks pp, 5 years of follow-up: number analyzed (Participants) | 21717
  > 14 weeks and ≤ 52 weeks pp, 5 years of follow-up | 4.55 [4.12 to 5.02]
  > 52 weeks pp or no delivery, 5 years of follow-up: number analyzed (Participants) | 228834
  > 52 weeks pp or no delivery, 5 years of follow-up | 4.88 [4.74 to 5.02]

25. Secondary Outcome: Adjusted Hazard Ratio (HR) for Postpartum Timing and IUD Expulsion-first Observed IUD Insertions
Description: Adjusted for propensity score and breastfeeding status, to evaluate whether the risk of IUD expulsion before and after 49 days of insertion among women who had a first observed IUD insertion within different time periods postpartum differs from the risk of IUD expulsion among women who had their first observed IUD insertion more than 52 weeks postpartum, including women without a recorded delivery within the past 52 weeks Reference group: IUD insertion > 52 weeks postpartum
Time Frame: Up to 11 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted hazard ratio
  Within 49 days, ≤ 6 weeks postpartum (pp): number analyzed (Participants) | 20060
  Within 49 days, ≤ 6 weeks postpartum (pp) | 1.93 [1.59 to 2.35]
  Within 49 days, > 6 weeks and ≤ 14 weeks pp: number analyzed (Participants) | 56047
  Within 49 days, > 6 weeks and ≤ 14 weeks pp | 0.88 [0.74 to 1.05]
  Within 49 days, > 14 weeks and ≤ 52 weeks pp: number analyzed (Participants) | 21717
  Within 49 days, > 14 weeks and ≤ 52 weeks pp | 1.38 [1.14 to 1.68]
  After 49 days, ≤ 6 weeks pp: number analyzed (Participants) | 20060
  After 49 days, ≤ 6 weeks pp | 1.32 [1.15 to 1.53]
  After 49 days, > 6 weeks and ≤ 14 weeks pp: number analyzed (Participants) | 56047
  After 49 days, > 6 weeks and ≤ 14 weeks pp | 1.03 [0.92 to 1.16]
  After 49 days, > 14 weeks and ≤ 52 weeks pp: number analyzed (Participants) | 21717
  After 49 days, > 14 weeks and ≤ 52 weeks pp | 1.39 [1.23 to 1.57]

26. Secondary Outcome: Adjusted Hazard Ratio (HR) for Postpartum Timing Risk 14-week Cut Point and IUD Expulsion-first Observed IUD Insertions
Description: Adjusted for propensity scores, to estimate the risk of IUD expulsion among women who had a first observed IUD insertion early in the postpartum period (i.e., up to 14 weeks postpartum) versus those who had a first observed IUD insertion late in the postpartum period (i.e., more than 14 weeks postpartum, including women without recorded delivery within the past 52 weeks). Reference group: IUD insertion >14 weeks postpartum or with no recorded delivery
Time Frame: Up to 11 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted hazard ratio | 0.88 [0.83 to 0.94]

27. Secondary Outcome: Adjusted Hazard Ratio (HR) for Postpartum Timing Risk 36-week Cut Point and IUD Expulsion-first Observed IUD Insertions
Description: Adjusted for propensity scores, to estimate the risk of IUD expulsion among women who had a first observed IUD insertion ≤ 36 weeks postpartum versus women who had a first observed IUD insertion > 36 weeks postpartum, including women without recorded delivery within the past 52 weeks. Reference group: IUD insertion >36 weeks postpartum or with no recorded delivery
Time Frame: Up to 11 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted hazard ratio | 0.95 [0.89 to 1.00]

28. Secondary Outcome: Adjusted Incidence Rate Ratio (IRR) for IUD Expulsion-first Observed IUD Insertions
Description: Overall and stratified by breastfeeding status at the time of IUD insertion for IUD expulsion for ≤ 36 weeks postpartum at IUD insertion versus > 36 weeks postpartum or with no recorded delivery, at 1 year and 5 years of follow-up Reference group: > 36 weeks or no delivery
Time Frame: At 1 year and 5 years of follow-up
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: adjusted incidence rate ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted incidence rate ratio
  Overall, 1 year of follow-up | 1.21 [1.12 to 1.30]
  Overall, 5 years of follow-up | 1.20 [1.13 to 1.28]
  Breastfeeding, 1 year of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 1 year of follow-up | 0.60 [0.44 to 0.85]
  Not breastfeeding, 1 year of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 1 year of follow-up | 1.25 [1.16 to 1.35]
  Breastfeeding, 5 years of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 5 years of follow-up | 0.80 [0.59 to 1.10]
  Not breastfeeding, 5 years of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 5 years of follow-up | 1.23 [1.15 to 1.31]

29. Secondary Outcome: Adjusted Incidence Rate Difference (IRD) for IUD Expulsion-first Observed IUD Insertions
Description: Adjusted incidence rate differences (per 1,000 person-years) for IUD expulsion for women ≤ 36 weeks postpartum at IUD insertion compared with those who were > 36 weeks postpartum or with no recorded delivery, 1 year of follow-up and 5 years of follow-up, overall and stratified by breastfeeding status Reference group: > 36 weeks or no delivery
Time Frame: At 1 year and 5 years of follow-up
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
per 1000 person-years
  Overall, 1 year of follow-up | 4.28 [2.50 to 6.06]
  Overall, 5 years of follow-up | 2.37 [1.53 to 3.22]
  Breastfeeding, 1 year of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 1 year of follow-up | -10.79 [-19.43 to -2.15]
  Breastfeeding, 5 years of follow-up: number analyzed (Participants) | 64186
  Breastfeeding, 5 years of follow-up | -2.62 [-6.51 to 1.26]
  Not breastfeeding, 1 year of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 1 year of follow-up | 5.11 [3.27 to 6.94]
  Not breastfeeding, 5 years of follow-up: number analyzed (Participants) | 30631
  Not breastfeeding, 5 years of follow-up | 2.65 [1.78 to 3.53]

30. Secondary Outcome: Crude Incidence Rate of IUD Expulsion Stratified by IUD Type-first Observed IUD Insertions
Description: as for outcome 1
Time Frame: Up to 11 years
Population: Women with either LNG-IUD (levonorgestrel-releasing intrauterine system) or copper IUD insertions
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 322898
per 1000 person-years
  LNG-IUD: number analyzed (Participants) | 259534
  LNG-IUD | 13.95 [13.63 to 14.28]
  Copper IUD: number analyzed (Participants) | 63664
  Copper IUD | 14.08 [13.44 to 14.75]

31. Secondary Outcome: Cumulative Incidence of IUD Expulsion Stratified by IUD Type-first Observed IUD Insertions
Description: as for outcome 2
Time Frame: At 1 year and 5 years of follow-up
Population: Women with either LNG-IUD (levonorgestrel-releasing intrauterine system) or copper IUD insertions
Measure: Number (95% Confidence Interval); unit: number of outcomes/IUD insertions (%)
Arm/Group | Women With IUD
Number analyzed (Participants) | 322898
number of outcomes/IUD insertions (%)
  LNG-IUD, 1 year of follow up: number analyzed (Participants) | 259234
  LNG-IUD, 1 year of follow up | 2.30 [2.24 to 2.36]
  Copper IUD, 1 year of follow up: number analyzed (Participants) | 63664
  Copper IUD, 1 year of follow up | 2.30 [2.18 to 2.44]
  LNG-IUD, 5 years of follow up: number analyzed (Participants) | 259234
  LNG-IUD, 5 years of follow up | 4.52 [4.40 to 4.65]
  Copper IUD, 5 years of follow up: number analyzed (Participants) | 63664
  Copper IUD, 5 years of follow up | 4.82 [4.56 to 5.10]

32. Secondary Outcome: Adjusted Hazard Ratio (HR) for IUD Type and IUD Expulsion-first Observed IUD Insertions
Description: Propensity score adjusted to evaluate whether the risk of IUD expulsion among women with LNG-releasing IUD at the time of first observed IUD insertion differs from the risk of IUD expulsion among women with copper IUD at the time of first observed IUD insertion
Time Frame: Up to 11 years
Population: Women with either LNG-IUD (levonorgestrel-releasing intrauterine system) or copper IUD insertions
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 322898
adjusted hazard ratio | 0.69 [0.65 to 0.73]

33. Secondary Outcome: Crude Incidence Rate of IUD Expulsion Stratified by Menorrhagia Status-first Observed IUD Insertions
Description: as for outcome 1
Time Frame: Up to 11 years
Population: Women with menorrhagia (heavy menstrual bleeding) status (yes/no) available in the 12 months before IUD insertion
Measure: Number (95% Confidence Interval); unit: per 1000 person-years
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
per 1000 person-years
  Yes: number analyzed (Participants) | 32552
  Yes | 39.56 [38.03 to 41.13]
  No: number analyzed (Participants) | 294106
  No | 11.10 [10.83 to 11.38]

34. Secondary Outcome: Cumulative Incidence of IUD Expulsion Stratified by Menorrhagia Status-first Observed IUD Insertions
Description: as for outcome 2
Time Frame: At 1 year and 5 years of follow-up
Population: Women with menorrhagia (heavy menstrual bleeding) status (yes/no) available in the 12 months before IUD insertion
Measure: Number (95% Confidence Interval); unit: number of outcomes/IUD insertions (%)
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
number of outcomes/IUD insertions (%)
  Yes, 1 year of follow-up: number analyzed (Participants) | 32552
  Yes, 1 year of follow-up | 6.89 [6.60 to 7.20]
  No, 1 year of follow-up: number analyzed (Participants) | 294106
  No, 1 year of follow-up | 1.78 [1.73 to 1.84]
  Yes, 5 years of follow-up: number analyzed (Participants) | 32552
  Yes, 5 years of follow-up | 11.89 [11.40 to 12.41]
  No, 5 years of follow-up: number analyzed (Participants) | 294106
  No, 5 years of follow-up | 3.72 [3.61 to 3.83]

35. Secondary Outcome: Adjusted Hazard Ratio (HR) for Menorrhagia Status and IUD Expulsion-first Observed IUD Insertions
Description: Propensity score adjusted to evaluate whether the risk of IUD expulsion among women using an IUD who have at least one diagnosis code indicating menorrhagia in the 12 months before IUD insertion differs from the risk of IUD expulsion among women who do not have this indication
Time Frame: Up to 11 years
Population: Women with menorrhagia (heavy menstrual bleeding) status (yes/no) available in the 12 months before IUD insertion
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
adjusted hazard ratio | 2.79 [2.62 to 2.98]

36. Secondary Outcome: Effect Modification of IUD Type on Breastfeeding Status for IUD Expulsion
Description: Propensity score-adjusted hazard ratios to evaluate the extent to which type of IUD (LNG-IUD vs. copper IUD) modified the association between IUD expulsion and breastfeeding among women who were and were not breastfeeding at the time of first observed IUD insertion
Time Frame: Up to 11 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 94205
adjusted hazard ratio
  LNG-IUD, breastfeeding yes vs.no: number analyzed (Participants) | 72201
  LNG-IUD, breastfeeding yes vs.no | 0.72 [0.64 to 0.80]
  Copper IUD, breastfeeding yes vs.no: number analyzed (Participants) | 22004
  Copper IUD, breastfeeding yes vs.no | 0.66 [0.54 to 0.80]

37. Secondary Outcome: Effect Modification of IUD Type on Postpartum Timing for IUD Expulsion
Description: Adjusted for propensity score and breastfeeding status, to evaluate the extent to which type of IUD (LNG-IUD vs. copper IUD) modified the association between IUD expulsion and postpartum timing of IUD insertion for women with IUD insertion at different time periods postpartum (i.e., ≤ 6 weeks, > 6 and ≤ 14 weeks, > 14 and ≤ 52 weeks) versus IUD insertion more than 52 weeks postpartum, including no recorded delivery within the past 52 weeks, at the time of the first observed IUD insertion. Reference group: LNG-IUD or Copper IUD, > 52 weeks or no delivery
Time Frame: Up to 11 years
Population: Women with either LNG-IUD (levonorgestrel-releasing intrauterine system) or copper IUD insertions
Measure: Number (95% Confidence Interval); unit: adjusted hazard ratio
Arm/Group | Women With IUD
Number analyzed (Participants) | 322898
adjusted hazard ratio
  LNG-IUD, ≤ 6 weeks: number analyzed (Participants) | 15631
  LNG-IUD, ≤ 6 weeks | 1.59 [1.38 to 1.82]
  LNG-IUD, > 6 to ≤ 14 weeks: number analyzed (Participants) | 42760
  LNG-IUD, > 6 to ≤ 14 weeks | 1.01 [0.90 to 1.14]
  LNG-IUD, > 14 to ≤ 52 weeks: number analyzed (Participants) | 16110
  LNG-IUD, > 14 to ≤ 52 weeks | 1.40 [1.23 to 1.58]
  Copper IUD, ≤ 6 weeks: number analyzed (Participants) | 4228
  Copper IUD, ≤ 6 weeks | 1.23 [0.98 to 1.53]
  Copper IUD, > 6 to ≤ 14 weeks: number analyzed (Participants) | 12934
  Copper IUD, > 6 to ≤ 14 weeks | 0.96 [0.81 to 1.13]
  Copper IUD, > 14 to ≤ 52 weeks: number analyzed (Participants) | 5379
  Copper IUD, > 14 to ≤ 52 weeks | 1.35 [1.13 to 1.63]

38. Secondary Outcome: Number of Indicators of a Potentially Difficult Insertion, Overall, by Breastfeeding Status, and by Postpartum Timing of IUD Insertion-first Observed IUD Insertions
Description: To describe the prevalence of indicators of a difficult IUD insertion (e.g., need for cervical dilation, ultrasound guidance, paracervical block, clinician not indicating difficulty, use of misoprostol among all users)
Time Frame: Up to 11 years
Population: Women with first observed IUD insertions
Measure: Number; unit: indicators
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
indicators
  Overall | 29777
  Breastfeeding: number analyzed (Participants) | 64186
  Breastfeeding | 1686
  Not breastfeeding: number analyzed (Participants) | 30631
  Not breastfeeding | 1077
  ≤ 6 weeks postpartum: number analyzed (Participants) | 20060
  ≤ 6 weeks postpartum | 573
  > 6 weeks and ≤ 14 weeks postpartum: number analyzed (Participants) | 56047
  > 6 weeks and ≤ 14 weeks postpartum | 1261
  > 14 weeks and ≤ 52 weeks postpartum: number analyzed (Participants) | 21717
  > 14 weeks and ≤ 52 weeks postpartum | 1146
  > 52 weeks postpartum or no delivery: number analyzed (Participants) | 228834
  > 52 weeks postpartum or no delivery | 26797

39. Secondary Outcome: Number of Indicators of a Potentially Difficult Insertion, Overall, by IUD Type and by Menorrhagia Status-first Observed IUD Insertions
Description: as for outcome 38
Time Frame: Up to 11 years
Population: Women with first observed IUD insertions
Measure: Number; unit: indicators
Arm/Group | Women With IUD
Number analyzed (Participants) | 326658
indicators
  Overall | 29777
  LNG-IUD: number analyzed (Participants) | 259234
  LNG-IUD | 24666
  Copper IUD: number analyzed (Participants) | 63664
  Copper IUD | 4648
  With menorrhagia in the past year: number analyzed (Participants) | 32552
  With menorrhagia in the past year | 3754
  Without menorrhagia in the past year: number analyzed (Participants) | 294106
  Without menorrhagia in the past year | 26023

ADVERSE EVENTS:
Time Frame: Retrospective analysis of data from 2001 to 2018
Description: This research study used secondary data from which personal identifiers were removed. The outcomes of uterine perforation and IUD expulsion are reported in the study results. Based on current guidelines from ISPE and the EMA, non-interventional studies conducted using electronic claims and health care records do not require reporting of adverse events or reactions
Arm/Group | Women With IUD
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall ensure that a written manuscript of any intended publication will be provided to BAYER at least 30 days prior to the intended submission or presentation in order to allow BAYER to review it. PI further agrees, upon written request from BAYER, not to submit such abstract or manuscript for publication or to make such presentation for the reasonably required time in order to allow for actions to be taken, which are necessary for BAYER to preserve rights to patents.

DOCUMENTS (2):
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT03754556/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03754556/SAP_001.pdf